CLINICAL TRIAL: NCT02893995
Title: A 16-Week, Open-Label, Multi-Center, Parallel, Randomized Controlled Study to Compare the Safety, Tolerability, Pharmacokinetics and Efficacy of Slow and Rapid Dose Titration Regimens of Subcutaneous Remodulin Therapy in Subjects With Pulmonary Arterial Hypertension
Brief Title: Safety, Tolerability, Pharmacokinetics and Efficacy of Two Different Rates of Subcutanous Remodulin® Dose Titration in Pulmonary Arterial Hypertension
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Business decision
Sponsor: United Therapeutics (Industry)
Collaborators: CVie Therapeutics Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CVT-CV-003
Record Dates: First submitted 2016-08-24; First posted 2016-09-09 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: PAH; Subcutaneous Treprostinil; Remodulin; 6 Minute Walk Test
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — treprostinil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Slow Dose Titration Group of Subcutaneous Treprostinil (Experimental): Remodulin (1.0, 2.5, 5 and 10 mg/ml formulations as available) will be administered by continuous subcutaneous infusion via a subcutaneous cannula using a microbore infusion tubing set and a micro infusion pump. While hospitalized, initiation will begin at approximately 1.25 ng/kg/min of subcutaneous treprostinil with dose increases of approximately 1.25 ng/kg/min once every seven days for the first 4 weeks, then approximately 2.5 ng/kg/min every seven days thereafter according to clinical response and tolerability.
  Interventions: Drug: Slow Dose Titration Group of Subcutaneous Treprostinil
- Rapid Dose Titration Group of Subcutaneous Treprostinil (Experimental): Remodulin (1.0, 2.5, 5 and 10 mg/ml formulations as available) will be administered by continuous subcutaneous infusion via a subcutaneous cannula using a microbore infusion tubing set and a micro infusion pump. While hospitalized, initiation will begin at approximately 2.0 ng/kg/min with dose increments of 1-2 ng/kg/min approximately every 12 hours according to clinical response and tolerability. Following subject discharge, the dose rate should be increased by 1-2 ng/kg/min with dose increments separated by at least 24 hours. When a dose rate of 20 ng/kg/min has been achieved the dose increments can be increased up to 4 ng/kg/min with dose increments separated by at least 24 hours. The aim is to achieve a dose rate of at least 10, 20, 30 and 40 ng/kg/min by the end of Weeks 1, 4, 8 and 12, respectively.
  Interventions: Drug: Rapid Dose Titration Group of Subcutaneous Treprostinil

INTERVENTIONS:
Drug: Slow Dose Titration Group of Subcutaneous Treprostinil — subcutaneous treprostinil
  Other Names: Remodulin
  Arms: Slow Dose Titration Group of Subcutaneous Treprostinil
Drug: Rapid Dose Titration Group of Subcutaneous Treprostinil — subcutaneous treprostinil
  Other Names: Remodulin
  Arms: Rapid Dose Titration Group of Subcutaneous Treprostinil

SUMMARY:
This is an open-label, multicenter, parallel, randomized (1:1 Slow Dose Titration Group; Rapid Dose Titration Group), two-group study to evaluate the safety, tolerability, pharmacokinetics and efficacy of slow and rapid dose titration regimens of subcutaneous Remodulin infusion in subjects with pulmonary arterial hypertension (PAH). The study will include about 50 subjects at up to 10 clinical trial centers in China. The treatment phase of the study will last approximately 16 weeks. Subjects who complete all required assessments will also be eligible to enter a long-term open-label, extension study (CVT-CV-004).

ELIGIBILITY:
Inclusion Criteria:

A subject is eligible for inclusion in this study if all of the following criteria apply:

1. The subject voluntarily gives written informed consent to participate in the study.
2. The subject is at least 18 years of age at screening.
3. The subject weighs a minimum of 40 kg with a body mass index less than 40 kg/m2 at screening.
4. The subject has a diagnosis of idiopathic or heritable PAH, PAH associated with repaired congenital systemic-to-pulmonary shunts (at least one year since repair with respect to the date of providing informed consent), or PAH associated with connective tissue diseases.
5. The subject must have a baseline 6MWD between 150 and 550 meters, inclusive, in the absence of a concurrent injury, illness (other than PAH or a PAH related condition), or other confounding factor that would prevent the accurate assessment of the subject's exercise capacity.
6. The subject is either treatment naïve or is receiving a PDE-5 inhibitor and/or an ERA for at least 60 days prior to screening and on a stable dose for at least 30 days prior to screening and is willing to remain on a PDE-5 inhibitor and/or an ERA at the same dose for the duration of the 16-week treatment phase.
7. The subject must be optimally treated with conventional pulmonary hypertension therapy (e.g., oral vasodilators, oxygen, digoxin, etc.) with no additions, discontinuations, or dose changes for at least 14 days prior to screening (excluding diuretics and anticoagulant dose adjustments).
8. The subject has undergone right heart catheterization during the screening period (or within 3 years before screening) and been documented to have a mean pulmonary artery pressure (PAPm) of greater than or equal to 25 mmHg, a pulmonary arterial wedge pressure (PAWP) of less than or equal to 15 mmHg, and pulmonary vascular resistance (PVR) of more than 3 Wood units.
9. The subject has undergone echocardiography within 7 days prior to randomisation with evidence of clinically normal left systolic and diastolic ventricular function, absence of any clinically significant left sided heart disease (e.g., mitral valve stenosis) and absence of unrepaired congenital heart disease. Subjects with clinically insignificant left ventricular diastolic dysfunction due to the effects of right ventricular overload (i.e., right ventricular hypertrophy and/or dilatation) will not be excluded.
10. The subject has a previous ventilation perfusion lung scan and/or high resolution computerized tomography scan of the chest and/or pulmonary angiography that are consistent with the diagnosis of PAH (e.g., low probability of pulmonary embolism; absence of major perfusion defects).
11. The subject has pulmonary function tests done within 9 months prior to or during the screening period with the following:

    1. Total lung capacity (TLC) is at least 60% (of predicted value)
    2. Forced expiratory volume in one second/forced vital capacity (FEV1/FVC) ratio is at least 50%
12. Sexually active women of childbearing potential must practice true abstinence from intercourse when it is in line with their preferred and usual lifestyle, or use two different forms of highly effective contraception. Medically acceptable forms of effective contraception include: (1) approved hormonal contraceptive (such as birth control pills), (2) barrier methods (such as a condom or diaphragm) used with a spermicide, (3) an intrauterine device (IUD), or (4) partner vasectomy. For women of childbearing potential, a negative serum pregnancy test is required at screening and a negative hCG urine pregnancy test is required at baseline visit. Women of child bearing potential include any females who have experienced menarche and who have not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation or bilateral oophorectomy) or are not postmenopausal (defined as amenorrhea for at least 12 consecutive months).

    Males participating in the study must use a condom during the length of the study, and for at least 48 hours after discontinuing study medication.
13. In the opinion of the Principal Investigator, the subject is able to communicate effectively with study personnel, is considered reliable, willing and likely to be cooperative with protocol requirements, including attending all study visits, and is mentally and physically capable of learning to administer Remodulin by continuous SC infusion using a micro infusion pump.

Exclusion Criteria:

A subject is not eligible for inclusion in this study if any of the following criteria apply:

1. The subject is pregnant or lactating.
2. The subject has received epoprostenol, treprostinil, iloprost or beraprost within 90 days prior to screening (except if used during acute vasoreactivity testing).
3. The subject has had previous intolerance or lack of efficacy to prostacyclin or a prostacyclin analogue that resulted in discontinuation or inability to titrate that therapy effectively.
4. The subject has any disease associated with PH other than idiopathic or heritable PAH, or PAH associated with repaired (for at least one year) congenital systemic-to-pulmonary shunts or connective tissue diseases or has had an atrial septostomy.
5. The subject is in WHO functional class IV.
6. The subject has a current diagnosis of uncontrolled sleep apnea as defined by their physician.
7. The subject has liver function tests (AST or ALT) greater than three times the upper limit of the laboratory reference range.
8. The subject has a history of active gastro-intestinal ulcer, intracranial hemorrhage, injury or other cause of clinically significant bleeding episode within 6 months before screening, or any other disease / condition that would either jeopardize the safety of the subject and / or interfere with the interpretation of study assessments in the opinion of the Investigator.
9. The subject has a history of ischemic heart disease including previous myocardial infarction or symptomatic coronary artery disease within 6 months before screening, or history of left sided myocardial disease as evidenced by a PAWP (or left ventricular end-diastolic pressure) greater than 15 mmHg or left ventricular ejection fraction (LVEF) less than 40%.
10. The subject has uncontrolled systemic hypertension as evidenced by systolic blood pressure greater than 160 mmHg or diastolic blood pressure greater than 100 mmHg.
11. The subject has systemic hypotension as evidenced by systolic blood pressure less than 85 mmHg
12. The subject has a musculoskeletal disorder (e.g., arthritis affecting the lower limbs, recent hip or knee joint replacement, artificial leg) or any other disease that is likely to limit ambulation, or is connected to a machine that is not portable.
13. The subject has an unstable psychiatric condition or is mentally incapable of understanding the objectives, nature, or consequences of the trial, or has any condition which in the Investigator's opinion would constitute an unacceptable risk to the subject's safety.
14. The subject is receiving an investigational drug, has an investigational device in place or has participated in an investigational drug or device study within 30 days prior to screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-02 (Estimated); Primary Completion 2018-04 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events Among Subjects through 16 Weeks | 16 Weeks
  The incidence of adverse events among subjects throughout the 16 week study will be measured by the number of subjects analyzed and the percentage of those subjects who experienced an adverse event.
Change in Patient Reported Site Pain from Baseline to Week 16 | Baseline and Week 16
  The site pain questionnaire is a 10-point scale rating the worst site pain experienced on a measured day. Scores will range from 0 (no pain) to 10 (worst possible pain). The questionnaire will be completed each time a new infusion site is placed and until a subject's infusion site pain level reaches a score of zero for two consecutive days or they have completed 14 days. Changes from Baseline to Week 16 will be summarized and compared between treatment groups using descriptive statistics. No formal hypothesis testing will be performed.
Incidence of Subject Discontinuations Among Participants through 16 Weeks | 16 Weeks
  The incidence of subject discontinuations among subjects throughout the 16 week study will be measured by the number of subjects analyzed and the percentage of those participants who discontinued.

SECONDARY OUTCOMES:
Change in 6-minute Walk Distance (6MWD) from Baseline to Week 16 | Baseline and Week 16
  The intent of the 6MWD test is to evaluate exercise capacity associated with carrying out activities of daily living. Change in 6MWD from Baseline to Week 16, correlates with the current clinical standard for assessing patient functional status in the treatment of PAH and is considered an objective measure of patient functional status by the American Thoracic Society (ATS). Subjects will be instructed to walk down a corridor at a comfortable speed as far as they could manage for six minutes. Distance <500 meters suggests considerable exercise limitation; Distance 500-800 meters suggests moderate limitation; Distance >800 meters (with no rests) suggests mild or no limitation. Changes from Baseline to Week 16 will be summarized and compared between treatment groups using descriptive statistics. No formal hypothesis testing will be performed.
Change in Borg Dyspnea Score (following 6MWT) from Baseline to Week 16 | Baseline and Week 16
  The Borg dyspnea score is a 10-point scale rating the maximum level of dyspnea (difficulty in breathing) experienced during the six-minute walk test (6MWT). The Borg dyspnea score will be assessed immediately following the 6MWT. Scores range from 0 (for no shortness of breath) to 10 (for the greatest shortness of breath ever experienced). Changes from Baseline to Week 16 will be summarized and compared between treatment groups using descriptive statistics. No formal hypothesis testing will be performed.
Change in N-terminal pro-B-type natriuretic peptide (NT-proBNP) concentrations from Baseline to Week 16 | Baseline and Week 16
  The N-terminal pro-BNP (NT-proBNP) serum concentration will be assessed as a biomarker to compare the severity of heart failure at Baseline and Week 16. Changes from Baseline to Week 16 will be summarized and compared between treatment groups using descriptive statistics. No formal hypothesis testing will be performed.
Number of Participants with a Change from Baseline World Health Organization (WHO) Functional Classification at Week 16 | Change from Baseline at Week 16
  The WHO Functional Class of pulmonary hypertension is a physical activity rating scale as follows: Class I: No limitation of physical activity. Class II: Slight limitation of physical activity. Class III: Marked limitation of physical activity. Class IV: Inability to carry out any physical activity without symptoms. Changes from Baseline to Week 16 will be summarized and compared between treatment groups using descriptive statistics. No formal hypothesis testing will be performed.
Change in PAH Symptoms from Baseline to Week 16 | Change from Baseline at 16 Weeks
  Symptoms of PAH including fatigue, dyspnea, edema, dizziness, syncope, chest pain and orthopnea will be assessed and if present, the intensity of the symptom will be rated as mild, moderate, or severe. Changes from Baseline to Week 16 will be summarized and compared between treatment groups using descriptive statistics. No formal hypothesis testing will be performed.
Change in Measured Tricuspid Annular Plane Systolic Excursion (TAPSE) from Baseline to Week 16 | Baseline and Week 16
  Change in right ventricular function will be assessed using the tricuspid annular plane systolic excursion (TAPSE) as determined by echocardiography. Changes from Baseline to Week 16 will be summarized and compared between treatment groups using descriptive statistics. No formal hypothesis testing will be performed.
Change in Measured Tricuspid Regurgitant Jet Velocity (TRJV) from Baseline to Week 16 | Baseline and Week 16
  Change in right ventricular function will be assessed using the tricuspid regurgitant jet velocity (TRJV) as determined by echocardiography. Changes from Baseline to Week 16 will be summarized and compared between treatment groups using descriptive statistics. No formal hypothesis testing will be performed.
Incidence of Pericardial Effusion from Baseline to Week 16 | Baseline and Week 16
  Change in right ventricular function will be assessed by the presence or absence of pericardial effusion as determined by echocardiography. Changes from Baseline to Week 16 will be summarized and compared between treatment groups using descriptive statistics. No formal hypothesis testing will be performed.
Measure treprostinil plasma concentration from Week 4 to Week 16 | Week 4, Week 8, Week 12, and Week 16
  During the treatment phase at Weeks 4, 8, 12, and 16 or at the time of premature study termination, a single blood sample will be collected to measure treprostinil plasma concentration.

CONTACTS AND LOCATIONS:
Overall Officials: Junbo Ge, Principal Investigator — Zhongshan Hospital affiliated with Fudan University
Locations (10):
- China (10):
  - Beijing Chao-Yang Hospital, Beijing
  - Beijing Anzhen Hospital, Capital Medical University, Beijing
  - Peking Union Medical College Hospital, Beijing
  - Fu Wai Hospital, Beijing
  - Beijing Shijitan Hospital, Beijing
  - Xiangya Hospital Centre South University, Changsha
  - Guangdong General Hospital, Guangzhou
  - Zhongshan Hospital affiliated with Fudan University, Shanghai
  - Shanghai Pulmonary Hospital, Shanghai
  - Wuhan Asia Heart Hospital, Wuhan